CLINICAL TRIAL: NCT02850718
Title: A Pivotal Study of the Bioequivalence of Oral Viagra® and a Test Sublingual Sildenafil Wafer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: iX Biopharma Ltd. (Other)
Collaborators: Linear Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SIL-003
Record Dates: First submitted 2016-04-12; First posted 2016-08-01 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Period 1: Sublingual wafer (Experimental): Subjects receive receive a single dose of 50 mg sublingual sildenafil followed by plasma sampling for 14 hours.
  Interventions: Drug: Sublingual Sildenafil
- Period 2: Oral comparator (Active Comparator): Subjects receive a single dose of 50 mg oral sildenafil (Viagra) followed by plasma sampling for 14 hours.
  Interventions: Drug: Oral Sildenafil

INTERVENTIONS:
Drug: Sublingual Sildenafil — 50 mg sildenafil sublingual wafer.
  Other Names: Pheonix
  Arms: Period 1: Sublingual wafer
Drug: Oral Sildenafil — 50 mg oral sildenafil (Viagra)
  Other Names: Viagra
  Arms: Period 2: Oral comparator

SUMMARY:
A comparative bioequivalence study in 48 healthy male volunteers of oral Viagra and a test sublingual sildenafil wafer.

DETAILED DESCRIPTION:
Healthy volunteers will complete two inpatient study periods and receive either sublingual wafer sildenafil or oral sildenafil. Plasma samples and adverse events will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily provides signed, written, and dated informed consent prior to any study-specific procedures.
2. Healthy male volunteers aged 18-50 years inclusive.
3. In good general health without clinically significant haematological, cardiac, respiratory, renal, endocrine, gastrointestinal, psychiatric, hepatic, or malignant disease, as determined by the Principal Investigator.
4. Sufficient access for venous cannulation to withdraw blood as per the study design.
5. Body mass index (BMI) of ≥19 to ≤ 30kg/m2 (inclusive).
6. Participant is deemed able to read and understand English in order to communicate with research staff and complete protocol required questionnaires and forms.
7. Able to refrain from smoking while at the research unit.

Exclusion Criteria:

1. Past history of hypersensitivity to sildenafil, any of its excipients, or severe allergic or anaphylactic reaction to any other drug.
2. A medical condition that, in the opinion of the Investigator, may adversely impact the participant's ability to complete the study, including but not limited to:

   1. History of priapism;
   2. History of easy fainting or symptomatic postural hypotension;
   3. Standing or supine systolic blood pressure < 90mmHg or diastolic blood pressure < 50mm Hg or postural drop of >30mm Hg;
   4. History of myocardial infarction or clinically significant cardiac disease including cardiac arrhythmia;
   5. History of retinitis pigmentosa or optic neuropathy or other risk factors of non-arteritic anterior ischaemic optic neuropathy (NAION);
   6. History or evidence of hypertension - defined as three BP readings (at rest) within 15 minutes of systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mmHg. Note: serial blood pressure readings are only required if the initial reading is elevated;
   7. Anaemia (haemoglobin < lower limit of normal for sex).
3. Clinically significant 12-lead ECG abnormalities at the screening visit as determined by the Investigator.
4. Concomitant consumption of any other medication regularly, with the exception of vitamins or minerals.
5. Consumption of drugs with either enzyme-inducing properties, such as rifampicin and St John's Wort, within 3 weeks prior to the initial dose of study drug and throughout the treatment phase or CYP3A4 inhibitors, such as erythromycin and clarithromycin, within 5 half-lives prior to the initial dose of study drug and throughout the treatment phase.
6. Previous known or suspected drug abuse (including analgesic drugs or tranquilizers) or dependence, as defined by DSM-IV, or history of alcohol abuse or excessive intake of alcohol, defined as regular weekly intake of >15 units for men and >10 units for women (1 unit= 25ml spirits,125ml wine, 250ml beer or lager).
7. Positive results on the urine drug screen indicative of illicit drug abuse or inconsistent with medication history, or alcohol breath test indicative of alcohol abuse.
8. History of hepatitis B or C, or other forms of non-infectious liver disease.
9. Clinically significant abnormalities in clinical chemistry, haematology, urinalysis, or serology results at screening that, in the opinion of the Investigator, puts the volunteer at risk for study participation.
10. Clinically significant plasma AST, ALT and ALP tests (defined as ≥1.5 times the upper limit of normal).
11. Positive serology for human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening.
12. Prevalent abnormality in the oral cavity which may alter sublingual drug absorption (e.g. recurrent oral ulceration, lichen planus, or xerostomia).
13. Any other condition which, in the opinion of the Investigator, makes the volunteer unsuitable for the study.
14. Unwillingness or inability to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the participant's ability to return for follow up visits on schedule.
15. Member or relative of study staff or the Sponsor directly involved in the study.
16. Previous participation in this study.
17. Has received another investigational agent or new chemical entity (defined as a compound which has not been approved for marketing) within 30 days prior to the Screening visit.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Sildenafil plasma concentrations | 1 week

SECONDARY OUTCOMES:
Number of patients with treatment-related adverse events | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Clinical Research, Perth, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No